CLINICAL TRIAL: NCT07012850
Title: Advanced Magnetic Resonance Imaging for Perioperative Evaluation of Dental, Oral and Maxillofacial Trauma
Status: Enrolling by invitation | Type: Observational
Sponsor: Harald Essig (Other)
Responsible Party: Sponsor-Investigator, Harald Essig, Prof. Dr. med. Dr. med. dent., University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: 2024-02307
Record Dates: First submitted 2025-05-09; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Traumatology; Maxillofacial Trauma; Maxillofacial Injuries
MeSH Terms: conditions — Maxillofacial Injuries | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — To reduce radiation exposure while simultaneously allowing for the visualization of soft tissues, newer imaging methods, including magnetic resonance imaging (MRI), as well as Black Bone and CT-like MRI protocols (ZTE, UTE), are being explored. These MRI techniques offer high-resolution, non-ionizing alternatives, showing promise for diagnosing soft tissue injuries and fractures without radiation risks.

SUMMARY:
Dental, oral, and maxillofacial trauma represents a significant public health concern, with most cases resulting from accidents and occurring frequently in young adults. Diagnosis relies on clinical examination and imaging modalities like computed tomography (CT) and cone-beam computed tomography (CBCT), which are standard for hard tissue assessment but expose patients to ionizing radiation. To reduce radiation exposure while simultaneously allowing for the visualization of soft tissues, newer imaging methods, including magnetic resonance imaging (MRI), as well as Black Bone and CT-like MRI protocols (ZTE, UTE), are being explored. These MRI techniques offer high-resolution, non-ionizing alternatives, showing promise for diagnosing soft tissue injuries and fractures without radiation risks, especially beneficial for younger patients. This study aims to assess MRI's diagnostic capabilities for maxillofacial trauma, focusing on early diagnosis, artifact reduction, and comparison to conventional X-ray-based imaging, within a minimal-risk study framework.

This study aims to evaluate the diagnostic efficacy of MRI compared to X-ray-based imaging modalities (CT/CBCT) for detecting dental, oral, and maxillofacial fractures, with a specific focus on Black Bone and CT-like MRI techniques. Additionally, it investigates MRI's potential to reduce artifacts around osteosynthesis plates, enhancing postoperative imaging quality in the presence of metal hardware.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with acute dental, oral and maxillofacial trauma
* Age: 18 years and older
* Able to give informed consent (documented by signature)
* No prior radiation-based imaging for the current trauma episode

Exclusion Criteria:

* Pregnant or lactating individuals
* Known contraindications to MRI (e.g., pacemakers, certain implants)
* Clinically significant concomitant diseases affecting imaging quality (e.g., severe neurocognitive disorders)
* Inability to comply with MRI procedures or study protocol (e.g., due to language barriers, psychological disorders, or dementia)
* Participation in other clinical trials that may interfere with the imaging study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study Population from the University Hospital Zurich, Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
qualitative imaging parameters | From enrollment to the end of treatment at week 5
  Primary Outcome Measures:
  1. Qualitative Assessment of Imaging Quality
  Description: Image quality will be evaluated using a standardized 5-point Likert scale for the following parameters: overall image quality, artifact severity, fracture visibility, and bone-to-soft-tissue contrast. Each parameter will be scored independently.
  Unit of Measure: Score on a 5-point Likert scale (1 = poor, 5 = excellent)
Quantitative Assessment of Fracture Dimensions | From enrollment to the end of treatment at week 5
  Fracture length, width, and depth will be measured in millimeters across axial, sagittal, and coronal planes using standardized digital radiologic tools. Measurements will be taken by two blinded radiologists and averaged.
  Unit of Measure: Millimeters (mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cranio-Maxillofacial and Oral Surgery, University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided